CLINICAL TRIAL: NCT06071143
Title: A Single Arm, Open-labelled, Dose-escalation, Single-center, Phase 1 Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Autologous Urine-derived Stem Cells, 『KDSTEM Inj.』, in Patients With Chronic Kidney Disease
Brief Title: Safety and Efficacy of KDSTEM Inj. in Patients With Chronic Kidney Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EHL Bio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KD-CP-22-1; 101473 (Other Grant/Funding Number: Republic of Korea Ministry of Food and Durg Safety)
Record Dates: First submitted 2023-10-03; First posted 2023-10-06 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Diseases
Keywords: CKD; Urine-derived Stem cell; stem cell; EHLBIO; UDSC
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KDSTEM Inj. (Experimental): 1. Low dose : Urine derived stem cells 1.0x10^8 cells
  2. High dose : Urine derived stem cells 3.0x10^8 cells
  Interventions: Biological: KDSTEM Inj.

INTERVENTIONS:
Biological: KDSTEM Inj. — 1. Low dose: The following study drugs are pre-mixed with 90mL of 0.9% normal saline and injected intravenously three times over the duration of the study. (Treatment group: KDSTEM Inj. 1.0x10^8 cells/10mL/2 syringes)
  2. High dose: The following study drugs are pre-mixed with 70mL of 0.9% normal saline and injected intravenously three times over the duration of the study. (Treatment group: KDSTEM Inj. 3.0x10^8 cells/30mL/6 syringes)

SUMMARY:
A Single arm, Open-labelled, Dose-escalation, Single-center, Phase 1 Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Autologous Urine-derived Stem Cells, 『KDSTEM Inj.』, in Patients with Chronic Kidney Disease.

The aim of this study is to evaluate the safety and preliminary efficacy of KDSTEM Inj. in the treatment in Patients with Chronic Kidney Disease.

DETAILED DESCRIPTION:
This clinical trial is a single-arm, open-labelled, dose-escalation, single-center Phase 1 study. Its aim is to evaluate the safety, tolerability, and preliminary efficacy of autologous urine-derived stem cells in patients with Chronic Kidney Disease.

If subjects voluntarily sign a written agreement to participate in this clinical trial, the subjects shall undergo the necessary examinations, as outlined in the clinical trial protocol, approximately one month prior to the administration of the investigational product.

After assessing the suitability of the subjects and ensuring participants meet the inclusion/exclusion criteria, eligible subjects will be assigned to different treatment arms. Subjects determined eligible by the investigator for receiving the investigational product on the scheduled administration day will receive a intravenous dose of the investigational product in visit 2, visit 3, and visit 4.

Safety and Efficacy assessments are conducted at 4, 8, 12, 16, 20, and 24 weeks after from the first administration to last administration of the investigational product, spanning a total of 24 weeks.

After all the subjects have completed visit 10, Safety and Efficacy will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 19 and 80 at the time of signing the agreement
2. Chronic kidney disease patients with an eGFR of 20 to 59 ml/min/1.73m² by MDRD at the screening and baseline
3. Male or female of childbearing age agreed to use accurate birth control method during this clinical trial
4. Subjects voluntarily signed an agreement in writing for this clinical trial

Exclusion Criteria:

1. Subjects who meet any of the following conditions at the screening visit

   1. Systemic infection
   2. HIV, HBV, HCV, Syphilis (+)
   3. Blood pressure higher than 190mmHg of SBP or 110mmHg of DBP
   4. AST or ALT higher than 3 times the upper limit of normal values
2. Subjects who received hemodialysis within 12 weeks prior to the screening or will be receive hemodialysis during this clinical trial
3. Subjects who received kidney transplantation or will be receive kidney transplantation during this clinical trial
4. Subjects diagnosed with the following diseases

   1. Solid Tumors or Hematologic Malignancies within 5 years prior to the screening
   2. Cognitive disorder, Alzheimer's disease or mental illness be clinically significant.
   3. Alcohol or drug abuse
   4. Severe Respiratory disease (Chronic Obstructive Pulmonary Disease, asthma, pneumonia, pulmonary embolism and pneumothorax, etc.)
   5. Stroke
   6. Heart related diseases (within 3 months prior to the screening severe cardiovascular conditions (angina Pectoris, myocardial infarction, unstable arrhythmia, heart failure, etc.)
5. Subjects who received cell therapy or another clinical trial product/device within 4 weeks prior to the screening
6. Subjects who were hypersensitivity reaction pertaining to penicillin, streptomycin, and amphotericin B
7. Subjects, as determined by an investigator, receiving treatment anticipated to affect the results of the clinical trials
8. Subjects being pregnant, providing breast milk, resulted in positive pregnancy test at screening or planning for pregnancy during this clinical trial
9. etc. Subjects determined unsuitable for this clinical trial by the investigator

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with treatment-related adverse events as assessed by CTCAE version 5.0 | 28 weeks follow-up after first injection
  vital sign, laboratory findings, physical exam, chest x-ray, cardiography, adverse drug reactions

SECONDARY OUTCOMES:
eGFR | From the first injection until 28 weeks later
  The variation in eGFR at each measurement compared to baseline measurement.
BUN | From the first injection until 28 weeks later
  The variation in BUN at each measurement compared to baseline measurement.
Serum creatinine | From the first injection until 28 weeks later
  The variation in Serum creatinine at each measurement compared to baseline measurement.
UPCR | From the first injection until 28 weeks later
  The variation and the rate of Change in UPCR at Each measurement compared to baseline measurement.
UACR | From the first injection until 28 weeks later
  The variation and the rate of Change in UACR at Each measurement compared to baseline measurement.
NGAL(Neutrophil Gelatinase Associated Lipocalin) | The first administration time, 4 weeks and 24 weeks after the third administration.
  Changes in NGAL (urine) and NGAL (plasma) at 4 weeks, 24 weeks measurement time after third injection compared to baseline
IL-6, IL-8, CCL18, TNF-α, α-Klotho | The first administration time, 4 weeks and 24 weeks after the third administration.
  Changes in IL-6, IL-8, CCL18, TNF-α, α-Klotho at 4 weeks, 24 weeks measurement time after third injection compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dae-Eun Choi, M.D, Ph.D, Principal Investigator — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, Chungcheongnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No